CLINICAL TRIAL: NCT02402114
Title: Hydrocortisone for Prevention of Post-Traumatic Stress Disorder
Acronym: HP-PTSD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Never started or submitted to IRB
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Principal Investigator, James Gardner, MD, Primary Investigator, Albert Einstein Healthcare Network
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HN4712
Record Dates: First submitted 2015-03-25; First posted 2015-03-30 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Post-Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Subject randomized to this group receives 1 oral dose of Hydrocortisone 120 mg
  Interventions: Drug: Hydrocortisone
- Placebo (Placebo Comparator): Subject randomized to this group will receive an oral sugar/placebo pill that looks similar to the Hydrocortisone pill.
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: Hydrocortisone — 120 mg Hydrocortisone given orally one time.
  Other Names: Cortef

SUMMARY:
Post-Traumatic Stress Disorder (PTSD) is an acquired psychiatric condition that occurs after exposure to a dangerous or life-threatening event. It is characterized by persistent fear- and stress-related symptoms, such as nightmares, flashbacks, depression, anxiety and guilt. These symptoms can interfere significantly with patients' lives and in some cases can be debilitating. One of the most frequent causes of PTSD is being a victim of a violent, interpersonal assault.

PTSD is felt to be primarily a disorder of memory formation - stressful memories are encoded too strongly in a patient's long-term memory, remaining too accessible and "present" to the patient long after the actual threat has passed. In recent years evidence has emerged that it may be possible to prevent PTSD by moderating the process of memory consolidation that occurs in the hours and days after a traumatic event.

Early research has suggested that enhancing the body's natural cortisol response to a stressful event may be a safe and effective way of moderating the process of memory consolidation and promoting adaptive, non-pathological memory encoding. In particular, the administration of hydrocortisone, a safe and widely used drug that mimics the body's own cortisol hormone, appears to reduce the risk of developing PTSD in patients who have sustained a traumatic event. However, this research is still in relatively early stages, and requires larger trials to confirm its efficacy. In addition, the research thus far has not adequately targeted assault victims, whom Investigator feel are some of the patients most likely to benefit from such an approach.

Investigators propose a prospective, placebo-controlled, double-blinded trial of administering single-dose oral hydrocortisone or placebo to 100 assault victims seen in the Einstein Medical Center Philadelphia Emergency Department to determine if this approach has efficacy in preventing PTSD. This study is designed as a pilot study, with the hopes that the data gathered in it can be used to design a larger and more robust trial in the future.

DETAILED DESCRIPTION:
Adult subjects will be screened in the Emergency Department (ED) by research associates. If they meet inclusion/exclusion criteria they will be offered enrollment. Subjects who choose to enroll will be randomized to receive either hydrocortisone 120mg PO, or placebo PO, one time in the Emergency Department. They will be given a packet of general information on traumatic stress and contact information for psychiatric assistance if they require it, but no further PTSD treatment will be given. Any further medical treatment will be at the discretion of the treating team.

At 6 weeks after enrollment subjects will be contacted by phone, and a brief structured interview, based on the PCL-S (a well-validated screening instrument for PTSD), will be administered by phone. Participants who screen positive will be informed that they may be suffering from PTSD, and will be offered the opportunity to seek care with the Einstein Psychiatry Department's PTSD program.

At 6 months after enrollment subjects will again be contacted and administered the PCL-C, as well as questions regarding other psychiatric comorbidities, substance use, and involvement in any further episodes of violence. In addition, review of subject medical records over the year since injury will be undertaken to determine if there is any difference in subsequent health-care utilization between those who received hydrocortisone vs placebo and between those who screen positive for PTSD vs those who don't.

ELIGIBILITY:
Inclusion Criteria:

1. Older than age 18
2. Presenting to ER for treatment of injuries sustained in a violent physical assault
3. Assault met DSM-IV "A" criterion (in patient's view, the assault involved or threatened death or serious injury)
4. Patient will be discharged home from Emergency Room

Exclusion Criteria:

1. Intoxicated due to drugs, alcohol or medication at the time they are approached.
2. Under arrest or in police custody at the time they are approached.
3. No memory of the assault
4. Cognitive impairment or psychosis identified by the treating physician or on chart review.
5. Patients whose presenting injury is a result of domestic (i.e. injured by a primary caregiver or significant other) or sexual violence
6. Under age 18
7. Not medically stable enough to participate
8. Non-English speakers
9. Pregnant or nursing women
10. Already on steroid treatment
11. Immunosuppressed (taking immunosuppressant medication, cancer undergoing active chemotherapy, AIDS, HIV not on HAART therapy)
12. Have an active infection identified by the treating physician or on chart review
13. Allergy or adverse reaction to hydrocortisone or other corticosteroids
14. Diabetic
15. On warfarin therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02-02 (Estimated); Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Positive PTSD screens | 6 weeks
  Percentage of patients that are PTSD positive on the PTSD Checklist scores (PCL-S) as per DSM-IV criteria after 6 weeks of enrollment

SECONDARY OUTCOMES:
Difference in PCL-S between HT group and placebo groups | 6 weeks
  Difference in PCL-S based on DSM VI criteria between HT group and placebo groups after 6 weeks of enrollment
Positive PTSD screens | 6 months
  Percentage of patients that are PTSD positive on the PTSD Checklist scores (PCL-S) as per DSM-IV criteria after 6 months of enrollment
Difference in PCL-S between HT group and placebo groups | 6 months
  Difference in PCL-S based on DSM VI criteria between HT group and placebo groups after 6 months of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: James Gardner, MD, Principal Investigator — Albert Einstein Healthcare Network
Locations (1):
- Albert Einstein Healthcare Network, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No